CLINICAL TRIAL: NCT02906085
Title: Investigations of the Endogenous Vasoconstrictor and Neuromodulator Peptide Endothelin-1 as a Potential Trigger of Migraine Aura
Brief Title: Endothelin-1 as a Potential Trigger of Migraine Aura
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Anders Hougaard, MD, PhD, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-16022143
Record Dates: First submitted 2016-09-03; First posted 2016-09-19 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Migraine With Aura
Keywords: [C10.228.140.546.399.750.250]
MeSH Terms: conditions — Migraine with Aura | interventions — Endothelin-1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endothelin-1 (Experimental): Intravenous infusion of pharmaceutical grade human endothelin-1
  Interventions: Drug: Endothelin-1
- Placebo (Placebo Comparator): Intravenous infusion of placebo (isotonic saline)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Endothelin-1
  Arms: Endothelin-1
Drug: Placebo — Isotonic saline
  Arms: Placebo

SUMMARY:
One third of migraine patients experience aura, i.e. dramatic, transient neurological symptoms, most often in the form of visual disturbances, that usually appear before the onset of migraine headache. The likely underlying mechanism of aura is known as cortical spreading depression, a wave of changes in electrical activity that slowly spreads in the outermost layer of the brain. It is currently not known what causes the aura to initiate in patients or what the relationship is between aura and migraine headache, e.g. if treatment targeted at aura mechanisms will prevent subsequent headache. Due to the short-lasting and unpredictable nature of aura, the only possible approach for systematic investigations is to experimentally trigger aura, but currently no method for aura-triggering is available.

The overall goal of the proposed project is to reveal the earliest mechanisms of the migraine attack by investigating the initiating factors of aura in the migraine brain.

Current animal evidence indicates that infusion of endothelin-1 (ET-1), a naturally occurring signaling molecule released from blood vessels, is safe and very likely to trigger migraine aura in patients.

In this project the investigators aim to study the effects of ET-1 on the human brain, to investigate aura-inducing effects of ET-1 in patients and to develop a safe and reliable method for the experimental induction of migraine aura using ET-1.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40 years
* Diagnosis of migraine with typical aura (patient group only)
* Attacks of migraine with aura at least once per month on average (patient group only)
* No history or family history of migraine (healthy subject group only)
* Use of safe contraception (women of fertile age only)

Exclusion Criteria:

* Tension-type headache more than one day per month on average
* Any other primary headache disorder
* Daily intake of medication
* Daily smoking during the past 5 years
* Pregnant or breastfeeding women
* Hypertension on the experimental day (systolic BP>150 mmHg or diastolic BP> 100 mmHg)
* History of any cardiovascular disease including cerebrovascular disease
* History of diabetes or hypercholesterolemia
* ECG changes suggestive of ischemia
* Contraindications of MRI

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of migraine aura | 0-24 hours

SECONDARY OUTCOMES:
Cerebral vasoconstriction: MR angiography | 0-30
  Time of flight arteriography using 3 tesla MRI (healthy subjects). Arterial diameters and circumferences (mm) will be measured from the resulting angiography images. This type of investigation will be carried out in healthy subjects only.
Change in cerebral blood flow: Phase contrast mapping | 0-30 minutes
  Cerebral blood flow (perfusion, ml/100 g/min) measured before and after intervention using MRI phase contrast mapping (measure of global brain perfusion). This type of investigation will be carried out in healthy subjects only.
Change in cerebral blood flow: Arterial spin labeling | 0-30 minutes
  Regional cerebral blood flow (perfusion, ml/100g/min) measured before and after intervention using MRI pseudo-continous arterial spin labelling at 3 tesla. This type of investigation will be carried out in healthy subjects only.

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Headache Center, Glostrup Municipality, Denmark